CLINICAL TRIAL: NCT05789992
Title: Detection of Nociceptive Stimulation and Anesthesia State by Equivalent Minimum Alveolar Concentration (eMAC) During Anesthesia With Varying Propofol and Remifentanil Concentrations
Brief Title: Evaluation of Equivalent Minimum Alveolar Concentration (eMAC) During Propofol/Remifentanil Anesthesia
Acronym: eMAC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhang Haopeng (Other)
Responsible Party: Sponsor-Investigator, Zhang Haopeng, Associate professor, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202302
Record Dates: First submitted 2023-03-02; First posted 2023-03-29 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: General Anaesthesia
MeSH Terms: interventions — Propofol; Intubation; Remifentanil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Group 1 BIS under tetanic electrical stimulation (Active Comparator): During tetanic electrical stimulation, and with propofol(random:3-5ug/ml) and remifentanil(random:0-3ng/ml), the response (body movement or hemodynamic change) was observed, and recorded it's BIS.
  Interventions: Drug: Propofol; Drug: Low Remifentanil; Procedure: tetanic electrical stimulation
- Group 2 eMAC under tetanic electrical stimulation (Active Comparator): During tetanic electrical stimulation or intubation, and with propofol(random:3-5ug/ml) and remifentanil(random:0-3ng/ml), the response (body movement or hemodynamic change) was observed, and recorded it's eMAC.
  Interventions: Drug: Propofol; Drug: Low Remifentanil; Procedure: tetanic electrical stimulation
- Group 3 BIS under intubation (Active Comparator): During intubation, and with propofol(random:3-5ug/ml) and remifentanil(random:3-5ng/ml), the response (body movement or hemodynamic change) was observed, and recorded it's BIS.
  Interventions: Drug: Propofol; Drug: Heigh Remifentanil; Procedure: Intubation
- Group 4 eMAC under intubation (Active Comparator): During intubation, and with propofol(random:3-5ug/ml) and remifentanil(random:3-5ng/ml), the response (body movement or hemodynamic change) was observed, and recorded it's eMAC.
  Interventions: Drug: Propofol; Drug: Heigh Remifentanil; Procedure: Intubation

INTERVENTIONS:
Drug: Propofol — Propofol (Random:3-5ug/ml)
  Other Names: Propofol for tetanic electrical stimulation and intubation
Drug: Low Remifentanil — Remifentanil (Random:0-3ug/ml)
  Other Names: Remifentanil for tetanic electrical stimulation
  Arms: Group 1 BIS under tetanic electrical stimulation; Group 2 eMAC under tetanic electrical stimulation
Drug: Heigh Remifentanil — Remifentanil (Random:3-5ug/ml)
  Other Names: Remifentanil for intubation
  Arms: Group 3 BIS under intubation; Group 4 eMAC under intubation
Procedure: Intubation — Endotracheal intubation before surgery
  Arms: Group 3 BIS under intubation; Group 4 eMAC under intubation
Procedure: tetanic electrical stimulation — tetanic electrical stimulation before surgery
  Arms: Group 1 BIS under tetanic electrical stimulation; Group 2 eMAC under tetanic electrical stimulation

SUMMARY:
The aim of this study is to verify the accuracy of eMAC compared to Bispectral Index (BIS) for depth and nociceptive stimulation monitoring of anesthesia during general anesthesia.

DETAILED DESCRIPTION:
eMAC is a new index based on response surface model for evaluating anesthesia state and anti-nociceptive stimulation levels. To valid it's clinical accuracy, a protocol was designed.

Patients will be allocated to receive a specific effect-site concentration of remifentanil and propofol during tonic electrical stimulation (5s, 50mA) and intubation. The concentration combinations include the electrical stimulation combination (effector chamber concentration random: remifentanil 0-3 ng/ml, propofol 3-5 ug/ml) and the intubation combination (effector chamber concentration random: remifentanil 3-5 ng/ml, propofol 3-5 ug/ml). All combinations were decided before operation. Every combination had a 5 min equilibration period, and the vital signs (Heart Rate, Blood pressure, any body movement) and BIS, eMAC will be recorded before and after the electrical stimulation and intubation. After this period, patients will be randomly allocated to receive an intravenous anesthesia or intravenous combined anesthesia, and regular anesthesia is executed. This study only records vital signs and BIS, eMAC during maintenance period of perioperative.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing elective surgery under general anesthesia;
2. Patients with ASA rating I~III;
3. The age of the patient is more than 18 years old;
4. The informed consent has been signed;

Exclusion Criteria:

1. Patients who are participating in other trials;
2. Patients with cognitive impairment, mental illness or taking psychotropic drugs within three months;
3. Patients with a history of stroke;
4. Patients with a history of alcoholism (long-term drinking more than 5 years, daily white wine consumption ≥ 50ml);
5. Pregnant women;
6. Patients with BMI>30;
7. Patients and family members who are unwilling to participate after understanding the research content;
8. According to the evaluation of the researcher, the actual condition is not suitable for the patients participating in this trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2023-04-29 (Actual); Study Completion 2023-04-29 (Actual)

PRIMARY OUTCOMES:
Prediction probability of eMAC | 1 year
  Prediction probability is an index(range:0-1) to describe the concordance between continuous measures and discrete scores. Prediction probability bettween eMAC and the lable of response was calculated.

SECONDARY OUTCOMES:
Prediction probability of BIS | 1 year
  Prediction probability is an index(range:0-1) to describe the concordance between continuous measures and discrete scores. Prediction probability bettween BIS and the lable of response was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Haopeng Zhang, Dr, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China

REFERENCES:
- [Background] Luginbuhl M, Schumacher PM, Vuilleumier P, Vereecke H, Heyse B, Bouillon TW, Struys MM. Noxious stimulation response index: a novel anesthetic state index based on hypnotic-opioid interaction. Anesthesiology. 2010 Apr;112(4):872-80. doi: 10.1097/ALN.0b013e3181d40368. PMID 20216387
- [Background] Gruenewald M, Ilies C, Herz J, Schoenherr T, Fudickar A, Hocker J, Bein B. Influence of nociceptive stimulation on analgesia nociception index (ANI) during propofol-remifentanil anaesthesia. Br J Anaesth. 2013 Jun;110(6):1024-30. doi: 10.1093/bja/aet019. Epub 2013 Mar 6. PMID 23471754
- [Background] Schumacher PM, Dossche J, Mortier EP, Luginbuehl M, Bouillon TW, Struys MM. Response surface modeling of the interaction between propofol and sevoflurane. Anesthesiology. 2009 Oct;111(4):790-804. doi: 10.1097/ALN.0b013e3181b799ef. PMID 19741484
- See also: For PubMed ID: 20216387 — https://pubs.asahq.org/anesthesiology/article/112/4/872/10694/Noxious-Stimulation-Response-IndexA-Novel
- See also: For PubMed ID: 19741484 — https://pubs.asahq.org/anesthesiology/article/111/4/790/9625/Response-Surface-Modeling-of-the-Interaction